CLINICAL TRIAL: NCT05094648
Title: Predictors of Success of High Flow Nasal Therapy in Covid 19 Patients
Brief Title: High Flow Nasal Therapy in Covid 19 Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maha Mahmoud Ahmed (Other)
Responsible Party: Sponsor-Investigator, Maha Mahmoud Ahmed, Assistant Lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: nasal therapy in covid patient
Record Dates: First submitted 2021-10-25; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: High Flow Nasal Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A: Covidpatient Who pass on high flow nasal therapy
  Interventions: Other: high flow nasal therapy
- group B: Covidpatient who failed on high flow nasal therapy and need NIV
  Interventions: Other: high flow nasal therapy

INTERVENTIONS:
Other: high flow nasal therapy — effect of high flow nasal therapy in covid 19 patients who pass and who need non invasive

SUMMARY:
This study aims to To identify factors that predict success of high flow nasal therapy in covid19 patients .

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) is a potentially fatal infection caused by the novel severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2)[1]. The highly contagious nature and exponential spread of SARS-CoV-2, coupled with its potential for a rapid progressto acute respiratory distress syndrome (ARDS), has overwhelmed health care systems globally, contributing to the high mortality rates in early reports [1,2].

The initial approach for respiratory support for severe COVID-19 pneumonia centredaround invasive mechanical ventilation and the standard lung protective strategy recommended for ARDS[3]. This may have been detrimental to a proportion of patients due to ventilator induced lung injury (VILI) and associated systemic inflammation[4]. Furthermore, other strategies to improve oxygenation may be more appropriate in patients with hypoxemic respiratory failure who do not require ventilatorysupport[4].

High-flow nasal oxygen (HFNO) is delivered by an air/oxygen blender, an active humidifier, a single heated circuit, and a nasal interface.

It delivers adequately heated and humidified medical gas at flow-rates of up to 60L/min, and is considered to have a number of physiological benefits, including the reduction of anatomical dead space and work of breathing, the provision of a constant fraction of inspired oxygen with adequate humidification and a degree of positive end-expiratory pressure (PEEP) [5,6].

ELIGIBILITY:
Inclusion Criteria:

* All Patients above 18 y old that will be diagnosed as COVID 19 based on PCR testing, who fulfil criteria that indicate need for high flow nasal therapy.

Exclusion Criteria:

* o Children less than 18 y old

  * Oropharyngeal and Nasopharyngeal swap negative patients
  * Patients who will refuse inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. demographic data including age, sex, smoking history, educational level.
  2. Duration of illness before admission, clinical presentation, presence of co morbidities, BMI.
  3. Vital signs, and radiologic findings
  4. ABG at admission and (half an hour, 2hr, 24 hr, and 48hr)later on.
  5. SPO2, FIO2, and respiratory rate at admission for calculating ROX index (SPO2/FIO2)/RR.
  6. GCC, and APACHI score at time of admission.
  7. Inflammatory markers at time of admission (CBC with differential, CRP, ferritin, D dimer, LDH), in addition to liver and renal function.
  At the end of the study patients will be claccifiedin to two groups based on success of high flow nasal therapy:
  Group A Covidpatient Who pass on high flow nasal therapy Group B Covidpatient who failed on nasal therapy and need NIV
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
predictors of success of high flow nasal therapy in covid 19 patients | Baseline
  This study aims to To identify factors that predict success of high flow nasal therapy in covid19 patients

REFERENCES:
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353